CLINICAL TRIAL: NCT05371873
Title: A Prospective Study of Early Warning and Predictive Indicators Related to the Individualized Staging and Prognosis in Liver Cancer Patients
Brief Title: A Study of Chromosomal Abnormalities as a Predictor of Staging and Prognosis in Patients With Liver Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, xiaqi, Director, First Affiliated Hospital of Zhejiang University
Other Study IDs: HCCpredictor
Record Dates: First submitted 2022-05-08; First posted 2022-05-12 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: microvascular invasion; minimal residual disease; circulating cell-free DNA; chromosomal abnormalities
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasm, Residual; Chromosome Aberrations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples were collected before and after liver resection, and tumor tissues were collected during surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anatomical resection group: Anatomical resection of liver cancer tissue
  Interventions: Procedure: Liver resection method
- Non-anatomical resection group: Non-anatomical resection of liver cancer tissue
  Interventions: Procedure: Liver resection method

INTERVENTIONS:
Procedure: Liver resection method — undergo anatomical or non-anatomical resection of liver cancer

SUMMARY:
Liver cancer is one of the most common malignant tumors worldwide with high morbidity and mortality, and hepatocellular carcinoma (HCC) is the main histological subtype. So far, liver resection is the most effective treatment but the postoperative recurrence rate is high at five years, and the prognosis is difficult to estimate. Microvascular invasion (MVI) and postoperative minimal residual disease (MRD) are crucial prognostic factors for patients undergoing hepatectomy. Although many laboratory and imaging methods have been established to estimate the recurrence risk, their stability and accuracy are still not high. To date, no unified conclusion is achieved. It's eagerly to screen out a batch of individualized staging and prognosis-related biological indicators for early warning and prediction of prognosis, having good stability and high precision. Circulating cell-free DNA (cfDNA) molecular detection technology is an emerging detection technology of tumor gene profiling in recent years, which can be used to predict and monitor tumor recurrence. In this study, by detecting genomic chromosomal abnormalities in plasma and tumor tissues of patients before and after surgery, the investigators hope to construct a preoperative MVI prediction model and a postoperative MRD monitoring model, so as to provide reference for the precise treatment of HCC.

DETAILED DESCRIPTION:
MVI and MRD confirmed by postoperative pathology are important prognostic factors for recurrence after liver resection, but current assessment methods have low sensitivity and specificity. cfDNA refers to the partially degraded endogenous DNA in the circulating blood that is free from the extracellular part of the body. When derived from dead and lysed tumor cells, it is called ctDNA, having a high chromosomal instability and relating to the tumor subtype and process. By low coverage whole genome sequencing, cfDNA and ctDNA in plasma were extracted and sequenced and chromosomal instability analysis is realized through UCAD pipeline. Therefore, the investigators can predict the trend of tumor by detecting cfDNA in patients, indicate MVI and MRD, carry out individualized staging of patients, predict recurrence and prognosis, and verify the prediction efficiency through follow-up, so as to establish corresponding prediction models.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years old;
* clinical diagnosis of liver cancer;
* intend to perform surgical treatment;
* postoperative pathological diagnosis of hepatocellular carcinoma;
* signed informed consent.

Exclusion Criteria:

* Not diagnosed with liver mass;
* Not undergo liver resection;
* Postoperative pathological diagnosis of non-hepatocellular carcinoma;
* Under the age of 18 or over 80;
* Concomitant pregnancy;
* Concomitant serious complications, including end-stage lung disease, unstable coronary heart disease or congestive heart failure grade 3-4, chronic kidney disease stage 4-5, cirrhosis (Child-Pugh) grade C, immunodeficiency;
* Incomplete data records.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators recruit patients dignosed with hepatocellular carcinoma without severe complications and other cancers. These patients eventually undergo liver resection.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
MVI model | 4 years
  Establish a preoperative prediction model of MVI by detecting chromosomal abnormalities in peripheral blood cfDNA
MRD monitor | 4 years
  Monitor postoperative MRD in postoperative patients and predict the recurrence risk and prognosis by detecting chromosomal abnormalities in peripheral blood cfDNA.

CONTACTS AND LOCATIONS:
Overall Officials: Min Zhang, director, Study Director — First Affiliated Hospital of Zhejiang University
Locations (1):
- The First Affiliated Hospital，College of Medicine，Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Heimbach JK, Kulik LM, Finn RS, Sirlin CB, Abecassis MM, Roberts LR, Zhu AX, Murad MH, Marrero JA. AASLD guidelines for the treatment of hepatocellular carcinoma. Hepatology. 2018 Jan;67(1):358-380. doi: 10.1002/hep.29086. No abstract available. PMID 28130846
- [Result] European Association for the Study of the Liver. EASL Clinical Practice Guidelines: Management of hepatocellular carcinoma. J Hepatol. 2018 Jul;69(1):182-236. doi: 10.1016/j.jhep.2018.03.019. Epub 2018 Apr 5. No abstract available. Erratum In: J Hepatol. 2019 Apr;70(4):817. doi: 10.1016/j.jhep.2019.01.020. PMID 29628281
- [Result] Imamura H, Matsuyama Y, Tanaka E, Ohkubo T, Hasegawa K, Miyagawa S, Sugawara Y, Minagawa M, Takayama T, Kawasaki S, Makuuchi M. Risk factors contributing to early and late phase intrahepatic recurrence of hepatocellular carcinoma after hepatectomy. J Hepatol. 2003 Feb;38(2):200-7. doi: 10.1016/s0168-8278(02)00360-4. PMID 12547409
- [Result] Pote N, Cauchy F, Albuquerque M, Voitot H, Belghiti J, Castera L, Puy H, Bedossa P, Paradis V. Performance of PIVKA-II for early hepatocellular carcinoma diagnosis and prediction of microvascular invasion. J Hepatol. 2015 Apr;62(4):848-54. doi: 10.1016/j.jhep.2014.11.005. Epub 2014 Nov 11. PMID 25450201
- [Result] Ye Q, Ling S, Zheng S, Xu X. Liquid biopsy in hepatocellular carcinoma: circulating tumor cells and circulating tumor DNA. Mol Cancer. 2019 Jul 3;18(1):114. doi: 10.1186/s12943-019-1043-x. PMID 31269959
- [Result] Wang D, Xu Y, Goldstein JB, Ye K, Hu X, Xiao L, Li L, Chang L, Guan Y, Long G, He Q, Yi X, Zhang J, Wang Z, Xia X, Zhou L. Preoperative evaluation of microvascular invasion with circulating tumour DNA in operable hepatocellular carcinoma. Liver Int. 2020 Aug;40(8):1997-2007. doi: 10.1111/liv.14463. Epub 2020 May 23. PMID 32279416
- [Derived] Shu Z, Ye T, Wu W, Su M, Wang J, Zhang M, Qian Z, Huang H, Zheng S, Xia Q. Preoperative plasma cell-free DNA chromosomal instability predicts microvascular invasion in hepatocellular carcinoma: a prospective study. BMC Cancer. 2025 May 13;25(1):867. doi: 10.1186/s12885-025-14268-9. PMID 40361115